CLINICAL TRIAL: NCT05480332
Title: Defining the Role of Endothelial Function Assessment Using EndoPAT in Cardiovascular Risk Screening : Comparison to Traditional Risk Assessment Tools and CIMT Testing
Status: Withdrawn | Type: Observational
Why Stopped: Unable to execute internal logistics
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Karthikeyan Ananthasubramaniam, MD, Henry Ford Health System
Other Study IDs: EndoPAT
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- EndoPAT Measured: Study participants who will undergo EndoPAT testing to obtain a non-invasive measurement of their endothelial function
  Interventions: Device: EndoPAT

INTERVENTIONS:
Device: EndoPAT — We will use the standard non-invasive EndoPAT finger probes to conduct the studies. A single finger on each hand will be placed into a probe equipped with pressure sensors. A baseline recording period will be obtained. After five minutes, an occlusion phase will start where a blood pressure cuff on the patient's non-dominant arm will be inflated to 60mmHg above the patient's systolic pressure, or 200mmHg, whichever is higher. This phase will be conducted in concert with the standard instructions provided with the EndoPAT system. The occlusion phase will last for five minutes, after which time the cuff will be deflated. There will then be a five minute post-occlusion recording period. The test will then be completed.
  The baseline period, occlusion period, and post-occlusion period will then be analyzed. A reactive hyperemia index score will be the desired output from the EndoPAT computer software, and will become the primary data point.

SUMMARY:
Our study aims to evaluate endothelial function using the non-invasive EndoPAT device, and compare this assessment to traditional cardiovascular risk calculation tools and carotid intima media thickness measurements. We look to determine whether the discovery of endothelial dysfunction provides incremental risk stratification over traditional and CIMT methods of cardiovascular risk assessment.

DETAILED DESCRIPTION:
Atherosclerosis is a disease affecting the function of arteries, and is one of the underlying causes of stroke, heart attack and other cardiovascular diseases. These diseases are some of the highest causes of morbidity and mortality in North America. As an inflammatory disease that involves the endothelium of blood vessels, atherosclerosis causes arteries to stiffen and become blocked with plaques. This leads to decreased function of these arteries, which at first is asymptomatic, but at later stages can block blood supply to the heart or brain.

The Endo-PAT 2000 is a device designed to measure endothelial function using finger probes placed onto the finger tip of a patient. It is made to detect the presence of peripheral endothelial dysfunction, which develops under the same mechanisms as coronary disease. Risk factors for heart disease are well recognized, and include gender, race, weight, smoking status, and the presence of hypertension, diabetes, and elevated cholesterol. While these factors are monitored in the clinical setting, the actual damage to vascular endothelium has previously been difficult to quantify. The EndoPAT system offers a novel method of assessing endothelial function as an aggregate outcome of all of these risk factors.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and older are eligible

Exclusion Criteria:

* None except age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients >/= 18 years consenting for participation are eligible. There are no speicifc exclusion critieria except age < 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05-01 (Estimated); Primary Completion 2016-05 (Estimated); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function as Indicated by the Reactive Hyperemia Index Score | Immediate